CLINICAL TRIAL: NCT05664945
Title: Rethinking Pulmonary Rehabilitation for Patients With COPD: a Three-arm Randomised Multicentre Trial (REPORT-trial)
Brief Title: Rethinking Pulmonary Rehabilitation - a Three-arm Randomised Multicentre Trial
Acronym: REPORT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Collaborators: University Hospital Bispebjerg and Frederiksberg (Other); Hillerod Hospital, Denmark (Other); Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Henrik Hansen, Principal Investigator, Copenhagen University Hospital, Hvidovre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-22015777
Record Dates: First submitted 2022-12-09; First posted 2022-12-27 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: A randomized clinical, assessor- and statistician blinded multicentre trial with three parallel-groups
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants will be informed that the trial is assessing the impact of pulmonary rehabilitation models on predetermined outcomes, but not the specific nature of the models of interest, and the predetermined hypothesis of the intervention group allocated to.
  All assessors are blinded to group allocation and previous test results. In case of failure keeping the outcome assessor blinded (that is, if a participant reveals his/her allocation) a second assessor will be available to step in and conduct the assessment on another day.
  To avoid investigators (subconscious) bias the biostatistician who perform the data analyses and validate the results is blinded to group allocation.
  The research group will interpret the results, before the allocation code is broken.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- pulmonary tele-rehabilitation (PTR) (Experimental): Recieve supervised PTR 2/weekly, session duration of 60 min; 35 min of exercise and 25min of patient education for 10-weeks (primary endpoint).
  Delivered from Hvidovre/Bispebjerg Hospital to groups of 4-6 patients who exercise at home and communicate via tablet-camera.
  After 10-weeks of PTR, participants are offered once weekly PTR for 60minuttes in groups of 4-8 patients throughout a 65-week maintenance period (secondary endpoint 75-weeks from baseline).
  Interventions: Behavioral: pulmonary tele-rehabilitation (PTR)
- home-based pulmonary rehabilitation (HPR) (Experimental): HPR is an individual self-initiated home-based PR program. Patient goal is to achieve at least 20 min of self-initiated muscle-endurance based exercise 3days/weekly for 10-weeks (primary endpoint).
  The first session is a home visit by an experienced respiratory physiotherapist and with focus on establishment of exercise goals, formal exercise prescription and education.
  The home visit is followed by 1/weekly session for 10-weeks.The sessions is delivered from Hvidovre/Bispebjerg Hospital via tablet-camera or telephone call.
  After 10-weeks of HPR, participants are offered once weekly PTR for 60min in groups of 4-8 patients throughout a 65-week maintenance period (secondary endpoint 75-weeks from baseline).
  Interventions: Behavioral: home-based pulmonary rehabilitation (HPR)
- Control (Active Comparator): Control group will receive usual care; medication, scheduled follow-up visit and possible phone contact with GP or the outpatient respiratory department. Except for assessment visits 10-, 35-, and 75-weeks from baseline no intervention is offered.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: pulmonary tele-rehabilitation (PTR) — PTR is delivered from promoter hospital to a group of 4-6 patients who exercise at home and communicate via tablet-camera.
  Each session is 60 min; 35 min exercise/ 25 min patient education, two times per week for a duration of 10-weeks (primary endpoint).
  Specific exercises are evidence-based; been used in several intervention studies on patients with COPD.
  Exercises involves larger muscle groups with 50/50 exercises for upper and lower extremities. Volume, intensity and content exercise protocol follow both national and international exercise recommendations.
  The education sessions consist of dialogue, reflections around empowerment and better living with COPD.
  Every fourth education session consists of 25 min Mindfulness exercises developed for COPD patients.
  After 10-weeks of PTR, participants are offered once weekly PTR for 60min in groups of 4-8 persons throughout a 65-week maintenance period (secondary endpoint 75-weeks from baseline).
  Arms: pulmonary tele-rehabilitation (PTR)
Behavioral: home-based pulmonary rehabilitation (HPR) — HPR is an individual self-initiated home-based PR aiming to achieve 20 min of self-initiated muscle-endurance based exercise; 3-days/weekly for 10-weeks (primary endpoint).
  Exercises are evidence-based; used in several intervention studies on patients with COPD and involves larger muscle groups with 50/50 exercises for upper/lower extremities.
  First session is a home visit by a respiratory physiotherapist. During the visit the physiotherapist and patient establish exercise goals, exercise prescription and provision of mindfulness exercises and educationbook.
  The home visit is followed by one weekly session for 10-weeks. A menu of topics relevant to COPD and self-management is discussed. A session is delivered from promoter hospital via tablet-camera or telephone call (patients' preference).
  After 10-weeks of HPR, participants are offered once weekly PTR for 60min in groups of 4-8 persons throughout a 65-week maintenance period (secondary endpoint 75-weeks from baseline).
  Arms: home-based pulmonary rehabilitation (HPR)
Behavioral: Control — Receive usual care; medication, scheduled follow-up visit and possible phone contact with GP and the outpatient respiratory department.
  Except for assessment visits 10-, 35-, and 75-weeks from baseline no intervention is offered.
  If a patient changes his/her mind and wishes to participate in a conventional hospital- or community-based PR program, it will be granted as this is a highly recommended treatment (e.g. rehabilitation after hospital admitted exacerbation).
  Arms: Control

SUMMARY:
Pulmonary rehabilitation (PR) is one of the cornerstones of care for people with COPD together with smoking cessation and medical treatment. Despite the compelling evidence for its benefits, pulmonary rehabilitation is delivered to less than 30% of patients with COPD. Access to PR are particularly challenging, and especially for those with the most progressed stages of the disease.

Pulmonary Tele-rehabilitation (PTR) and Home-based pulmonary rehabilitation (HPR) are two emerging models using health-care supportive technology that have proven equivalent to the conventional PR programs in patients with COPD who are able and willing to participate in conventional PR.

However, much remain unknown regarding patients with COPD unable to access and participate in the conventional out-patient hospital- or community-based PR when offered during routine consultation. No studies have been conducted to specifically intervene towards this group. Response from emerging rehabilitation models for this specific group is a black box with no substantial research.

To fulfill its potential of relevance, results from emerging models, such as Pulmonary Telerehabilitation and Home-based pulmonary rehabilitation must be of clinical relevance, and superior to the current 'usual care' (medication and scheduled follow-up control) in patients with COPD unable to access and participate in the conventional out-patient hospital- or community-based PR when offered during routine consultation.

DETAILED DESCRIPTION:
This trial will investigate if pulmonary tele-rehabilitation (PTR) and home-based pulmonary rehabilitation (HPR) leads to respiratory symptom relief (CAT score) and improvements on secondary outcomes in patients unable to access conventional rehabilitation programs (standard PR offer).

Our hypotheses in a three-arm RCT design are

1. PTR and HPR will be equivalent to each other
2. PTR and HPR will be superior to usual care, that is the control group (CON - no intervention)

ELIGIBILITY:
Inclusion Criteria:

* Indication for pulmonary rehabilitation according to Danish national guidelines
* Unable to access and participate in the conventional out-patient hospital- or community-based PR when offered during routine consultation
* A post-bronchodilator ratio FEV1/FVC <70% (confirmed physician diagnosis of COPD)
* A post-bronchodilator FEV1 <80% (degree of airway obstruction) corresponding to GOLD grade 2-4 (moderate to very severe)
* GOLD group B, C, D corresponding to severe respiratory symptoms and/or frequent acute exacerbations
* Able to stand up from a chair (height 44-46cm) and walk 10 meters independently (with or without a walking aid)
* Able to lift both arms to a horizontal level with a minimum of 1 kilogram's dumbbells in each hand

Exclusion Criteria:

* Participation in conventional PR in the past 24 months
* Cognitive impairment - unable to follow instructions
* Impaired hearing or vision - unable to see or hear instruction from a tablet
* Unable to understand and speak Danish
* Comorbidities where the exercise content is contraindicated (e.g. treatment for diabetic foot ulcer, active cancer treatment, life expectancy <12-months)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in COPD Assessment Test (CAT) | Baseline; 10-weeks from baseline (primary endpoint); 35-weeks from baseline; 75-weeks from baseline (secondary endpoint)
  Patient completed questionnaires that assess respiratory symptoms. Eight item questionaire with total score from 0-40 points.

SECONDARY OUTCOMES:
Change in 1-minute sit-to-stand test (1-min-STS) | Baseline; 10-weeks from baseline (primary endpoint); 35-weeks from baseline; 75-weeks from baseline (secondary endpoint)
  measures endurance
Change in 30seconds sit-to-stand test (30sec-STS) | Baseline; 10-weeks from baseline (primary endpoint); 35-weeks from baseline; 75-weeks from baseline (secondary endpoint)
  measures muscle strength
Change in Short Physcial Performance Battery (SPPB) | Baseline; 10-weeks from baseline (primary endpoint); 35-weeks from baseline; 75-weeks from baseline (secondary endpoint)
  Measures frailty/possible sarcopenia/ mobility disaabilities
Change in Handgrip strength (JAMAR) | Baseline; 10-weeks from baseline (primary endpoint); 35-weeks from baseline; 75-weeks from baseline (secondary endpoint)
  measures handgrip muscle strength in kilo. High is better
Changes in objectively measured physical acitivity (50% of total sample) | Baseline; 10-weeks from baseline ( primary endpoint); 35-weeks from baseline; 75-weeks from baseline (secondary endpoint)
  Devise is ActivePAL triaxial accelerometer (PAL Technologies Ltd., Glascow, UK). Wearing time is 24 h per day for 5 days at each time point. Measures sedentary and active body movements, steps per day and METs. High number of activity is better
Change in Hospital Anxiety and Depression Scale (HADS) | Baseline; 10-weeks from baseline (primary endpoint); 35-weeks from baseline; 75-weeks from baseline (secondary endpoint)
  Patient completed questionnaires that assess anxiety and depression symptoms. Seven item domain questions for depression with total score form 0-21 point. Seven item domain questions for anxiety with total score fra 0-21 points.
Change in Euro Qol (EQ5D-3L) | Baseline; 10-weeks from baseline (primary endpoint); 35-weeks from baseline; 75-weeks from baseline (secondary endpoint)
  Patient completed questionnaires that assess quality of life. Total score fra 0-1 on EQ5D-health domain. Total score from 0-100mm on EQ5D-vas domain. No total domain score
Change Brief Pain Inventory (BPI) | Baseline; 10-weeks from baseline (primary endpoint); 35-weeks from baseline; 75-weeks from baseline (secondary endpoint)
  Patient completed questionnaires that assess pain. Low score is better
Change Multidimensional Fatigue Inventory (MFI-20) | Baseline; 10-weeks from baseline (primary endpoint); 35-weeks from baseline; 75-weeks from baseline (secondary endpoint)
  Patient completed questionnaires that assess pain. Low score is better
Change Pittsburg Sleep Quality Index (PSQI) | Baseline; 10-weeks from baseline (primary endpoint); 35-weeks from baseline; 75-weeks from baseline (secondary endpoint)
  Interview completed questionnaire that assess sleep quality. Low score is better
Program completion | at 10-weeks from baseline (primary endpoint); 75-weeks from baseline (secondary endpoint)
  The number of participants who complete their allocated rehabilitation program (attend at least 70% of planned sessions).
Number of hospital admissions (respiratory related and all-cause) | at 10-weeks from baseline (primary endpoint); 35-weeks from baseline; 75-weeks from baseline (secondary endpoint)
  Total number
Mortality (respiratory related and all-cause) | at 10-weeks from baseline (primary endpoint); 35-weeks from baseline; 75-weeks from baseline (secondary endpoint)
  Total number
Adverse events | at 10-weeks from baseline (primary endpoint); 35-weeks from baseline; 75-weeks from baseline (secondary endpoint)
  numbers of SAE and AE

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Hansen, PhD, Principal Investigator — Dept. of Respiratory Medicine, University Hospital Hvidovre; Nina Godtfredsen, MD, PhD, Study Chair — Dept. of Respiratory Medicine, University Hospital Hvidovre
Locations (7):
- Denmark (7):
  - Copenhagen University Hospital Amager, Copenhagen, Greater Copenhagen
  - Copenhagen University Hospital Bispebjerg-Frederiksberg, Copenhagen, Greater Copenhagen
  - Copenhagen University Hospital Herlve-Gentofte, Gentofte Municipality, Greater Copenhagen
  - Copenhagen University Hospital Nordsjaelland, Hillerød, Greater Copenhagen
  - Copenhagen University Hospital Hvidovre, Hvidovre, Greater Copenhagen
  - Municipality of Copenhagen, Copenhagen
  - Bornholms Hospital, Rønne

IPD SHARING:
Plan to Share IPD: No
Access demands a part application to; (1) Danish Data Protection agency, (2) ethics committee of the capital region, (3) national health Data authorities.
  Only if the applications are approved data will be considered available for sharing. The investigator will not be able to support this process.

REFERENCES:
- [Background] Nielsen C, Godtfredsen N, Molsted S, Ulrik C, Kallemose T, Hansen H. Supervised pulmonary tele-rehabilitation and individualized home-based pulmonary rehabilitation for patients with COPD, unable to participate in center-based programs. The protocol for a multicenter randomized controlled trial - the REPORT study. PLoS One. 2025 Jan 7;20(1):e0312742. doi: 10.1371/journal.pone.0312742. eCollection 2025. PMID 39774509